CLINICAL TRIAL: NCT02111499
Title: A Randomized, Controlled, Observer-blind Psoriasis Plaque Test to Investigate the Anti-psoriatic Efficacy, Tolerability and Safety (Skin Atrophy) of LAS41004 Formulations in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: Efficacy, Tolerability and Safety of LAS41004 Formulations in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H553000-1308; 2013-003754-24 (EudraCT Number)
Record Dates: First submitted 2014-03-24; First posted 2014-04-11 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis
Keywords: psoriasis plaque test; topical application; atrophy measure
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- formulation 1 (Experimental): topical treatment, once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5
- formulation 2 (Experimental): topical treatment, once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5
- formulation 3 (Experimental): topical treatment, once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5
- formulation 4 (Experimental): topical treatment,once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5
- formulation 5 (Placebo Comparator): topical treatment, once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5
- formulation 6 (Active Comparator): topical treatment, once daily for 4 weeks
  Interventions: Drug: LAS41004-IMP1; Drug: LAS41004 IMP2; Drug: LAS41004 IMP3; Drug: LAS41004 IMP4; Drug: LAS41004 IMP6; Drug: LAS41004 IMP5

INTERVENTIONS:
Drug: LAS41004-IMP1 — daily topical application
Drug: LAS41004 IMP2 — daily topical application
Drug: LAS41004 IMP3 — daily topical application
Drug: LAS41004 IMP4 — daily topical application
Drug: LAS41004 IMP6 — daily topical application
Drug: LAS41004 IMP5 — once daily, topical

SUMMARY:
Clinical investigation of anti-psoriatic efficacy and atrophy

DETAILED DESCRIPTION:
In this trial three concentrations of bexarotene in combination with a fixed concentration of betamethasone dipropionate, as well as monotherapy with bexarotene, will be investigated regarding their efficacy, tolerability and safety in patients with mild to moderate plaque psoriasis and will be compared with the vehicle and an active comparator.

Since a side effect of the application of corticosteroids is skin atrophy, additionally three non-lesional test areas (not affected by psoriasis) on the volar forearm will be treated with the active reference product, one of the fixed combinations and the vehicle. Skin atrophy will be investigated by visual assessment and ultrasound at these test areas

ELIGIBILITY:
Main Inclusion Criteria:

* 18 to 75 years of age
* Men and women with skin type I to IV (Fitzpatrick 1974).
* Suffering from mild to moderate plaque psoriasis of at least 6 months duration that is amenable to local therapy.
* With at least one stable psoriatic plaque in an area sufficient for product application meeting the following criteria:

  * Located at the trunk and/or the extremities (plaques located on the head, palms, or soles of the feet, intertriginous or genitoanal areas are not suitable).
  * Plaques with a clinical score of the parameter erythema and or induration of ≥ 2 for each sign at the screening visit. At Day 1 each parameter has to be scored ≥ 2.
  * Where more than one plaque is to be used, plaques should be comparable, with at least "2" in each score for erythema and induration.
  * • Body surface area (BSA) involvement < 10 %.
* Prepared to give written informed consent specific to the trial, before any assessment is performed.
* • In the case of women of childbearing potential using reliable methods of contraception which result in a low failure rate i.e. less than 1% per year (e.g. contraceptive implants or injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner). During the study an additional barrier method (e.g. condoms) should be used. Non-childbearing potential is defined as surgical sterilization (hysterectomy, ovariectomy or tubal ligation), postmenopausal status (continuous amenorrhea of at least 2 years).
* In the case of men with partners of childbearing potential willingness of using condoms during the study conduct and 1 month after end of treatment.

Main Exclusion Criteria:

* • Patients who need systemic treatment for their psoriasis.

  * Severe forms of psoriasis or forms of psoriasis other than chronic plaque psoriasis,
  * Systemic treatment (see table below):

Corticosteroids, antibiotics 4 weeks prior to trial Day 1 and during conduct of trial Retinoids Ciclosporin Methotrexate Fumaric acid esters 3 months prior to trial Day 1 and during conduct of trial Anti-inflammatory substances, NSAIDs 2 weeks prior to trial Day 1 and during conduct of trial Biologics 6 months prior to trial Day 1 and during conduct of trial

* Topical treatment of all other body regions with corticosteroids or immunosuppressants where more than 20 % of the body surface area is treated.
* Diseases:

Significant skin infections caused by bacteria, viruses or fungi, including but not limited to tuberculosis, syphilis or varicella zoster infection Parasitic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve, AUC, of the width of the echo-lucent band based on sonography measurements | day 1 vs day 29
  The primary objective is to gain evidence suggesting efficacy of the investigational products in the treatment of plaque-type psoriasis as assessed by the AUC of the width of the echo-lucent band

SECONDARY OUTCOMES:
erythema and induration | day 1 vs day 29
  investigation of the individual scores for erythema and induration
local skin tolerability | every day for 28 days
  Safety investigation of tolerability parameters assessed by a dermatologist
atrophy | day1 vs day 29
  investigation of skin atrophy assessments on non-lesional test areas
assessment of (serious) Adverse Events | from baseline to day 29
  Daily record will be performed and - if needed - causality and severity assessed

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Dr med, Principal Investigator — proDERM GmbH
Locations (1):
- proDERM GmbH, Schenefeld, Schleswig-Holstein, Germany